CLINICAL TRIAL: NCT01956149
Title: Multicentre, Phase II Study With Cabazitaxel in Previously Treated Patients With Advanced or Metastatic Adenocarcinoma of the Oesophagogastric Junction and Stomach
Brief Title: Study With Cabazitaxel in Previously Treated Patients With Advanced or Metastatic Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CabaGast
Record Dates: First submitted 2013-07-03; First posted 2013-10-08 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-01

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; second-line treatment; Cabazitaxel; response
MeSH Terms: conditions — Stomach Neoplasms | interventions — cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cabazitaxel (Experimental): Cabazitaxel 20 mg/m2 over 1 hour i.v., repeated on day 22
  Interventions: Drug: Cabazitaxel

INTERVENTIONS:
Drug: Cabazitaxel — 20 mg/m2 over 1 hour i.v., repeated on day 22 for maximum 6 cycles.

SUMMARY:
Single-arm study to determine disease control rate in second- (or later) line treatment with cabazitaxel after the failure of palliative primary treatment.

DETAILED DESCRIPTION:
65 patients with advanced or metastatic adenocarcinoma of the oesophagogastric junction and stomach will be treated with 20mg/m2 Cabazitaxel for a maximum of 6 cycles. Main objective of the study is the Disease Control Rate (DCR) with Cabazitaxel.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed inoperable and/or metastatic adenocarcinoma of the oesophagogastric junction or stomach
2. Progression of a measurable lesion (RECIST) on previous palliative chemotherapy. Neoadjuvant/adjuvant treatment is not counted, unless progression occurs < 6 months after completion of the treatment. In these cases, neoadjuvant/adjuvant treatment is counted as one line.
3. Male and female patients aged > 18 years
4. ECOG ≤ 1
5. neutrophils ≥ 1500/µl
6. Haemoglobin ≥ 9 g/dl
7. Platelets ≥ 100,000/µl
8. AST/SGOT and/or ALT/SGPT ≤2.5 x ULN;
9. Total bilirubin ≤1.0 x ULN
10. Serum creatinine ≤ 1.5 times the normal value, or creatinine clearance ≥ 60 ml/min
11. Written patient informed consent

Exclusion Criteria:

1. A history of severe hypersensitivity to taxanes (≥ grade 3) or to medicinal products containing polysorbate 80 (≥ grade 3)
2. Active CAD, cardiomyopathy or NYHA stage III-IV heart failure
3. Malignant secondary disease dating back < 5 years (exceptions: in situ cervical carcinoma, appropriately treated basal cell carcinoma of the skin)
4. Severe secondary internal diseases, including uncontrolled diabetes mellitus or an acute infection
5. Concomitant medication or planned treatment with strong CYP450 3A4/5 inducers or inhibitors (list of medicinal products in the appendix) or the relevant medicinal products were not discontinued a minimum of one week before treatment
6. Peripheral polyneuropathy > NCI grade II
7. Severe hepatic impairment (AST/ALT > 2.5 x ULN, , bilirubin > 1 x ULN)
8. Chronic inflammatory bowel disease
9. Participation in another study
10. Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-09; Primary Completion 2017-12 (Actual); Study Completion 2018-04-04 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) | up to 17 months
  Patients are staged every 6 weeks during therapy (after cycle 2, 4 and 6, i.e. up to 18 weeks) and during follow-up (up to 12 months)

SECONDARY OUTCOMES:
Overall survival (OS) | up to 17 months
  From date of randomization until the date of death from any cause, assessed up to 17 months
Progression-free survival (PFS) | up to 17 months
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 17 months
Response rate by subgroup (with and without previous treatment with a taxane) | up to 17 months
  Patients are staged every 6 weeks during therapy (after cycle 2, 4 and 6, i.e. up to 18 weeks) and during follow-up (up to 12 months)
Toxicity | up to 18 weeks
  incidence and intensity of adverse events
Correlation of circulating tumor cells with PFS and OS | up to 18 weeks
  samples for analysis of circulating tumor cells are taken before therapy, before every new cycle, and at the end of treatment (every 3 weeks).
Correlation of circulating tumor cells with the clinical response | up to 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Harald Schmalenberg, MD, Principal Investigator — Krankenhaus Dresden Friedrichstadt
Locations (3):
- Germany (3):
  - Krankenhaus Dresden Friedrichstadt, Dresden
  - Krankenhaus Nordwest, Frankfurt am Main
  - Universitätsklinikum Jena, Jena